CLINICAL TRIAL: NCT00074763
Title: Randomized Crossover Study Comparing Fresh Random Platelets and Autologous Cryopreserved Thrombosol Treated Autologous Platelets
Brief Title: Comparing Fresh Random Platelets and Autologous Cryopreserved Thrombosol Treated Autologous Platelets
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to low recruitment.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0088
Record Dates: First submitted 2003-12-19; First posted 2003-12-23 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; ALL; CLL; AML; CML; MDS; Remission; Hematologic Disorder; Transfusion; Thrombosol; Autologous Platelet Transfusion; Platelet Transfusion; Single donor platelet apheresis; Cryopreservation; Thrombocytopenia
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Diseases; Thrombocytopenia | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet Transfusion (Experimental): ThromboSol-preserved autologous platelet transfusion or Standard platelet transfusion. All patients receive both platelets frozen with Thrombosol and fresh random platelets. The order in which patients receive these two types of platelets randomized in a crossover design. Patients randomly assigned to receive either the sequence FRP then Thrombosol or Thrombosol then FRP. The randomization will occur after second cycle of chemotherapy, since all patients will receive FRP with the first cycle.
  Interventions: Biological: Platelet Transfusion

INTERVENTIONS:
Biological: Platelet Transfusion — All receive both platelets frozen with Thrombosol and fresh random platelets (FRP), order received is randomized, i.e. receive either FRP then Thrombosol or Thrombosol then FRP.

SUMMARY:
Objectives:

* Determine the corrected count increment of autologous transfused platelets that had been stored by cryopreservation with ThromboSol.
* Determine the ability of autologous platelets that had been stored by cryopreservation with ThromboSol to correct thrombocytopenia.

DETAILED DESCRIPTION:
Platelets are an important component of blood. Transfusions with platelets help to control bleeding in thrombocytopenic patients. Using the standard blood banking procedures, platelets can only be stored for up to 5 days. This is to help decrease the risk of contamination with bacteria. Currently, it is not possible to use cryopreserved (frozen) platelets because the platelets are damaged during the freezing process. Therefore, long-term banking of platelets or autologous donation (storing your own platelets to be given back to you at a later time) has not been possible. ThromboSol is a new solution that was designed to allow platelets to be frozen without damaging them. The use of ThromboSol may allow for long-term banking of platelets and/or autologous donations.

During a period of cancer remission and when you have enough platelets in your blood, you will undergo an apheresis procedure to collect platelets. This procedure is similar to donating plasma to a blood bank. You will have up to 6 apheresis procedures (on different days) to collect up to 6 units of autologous platelets that can be transfused back to you. The platelets that are collected will be frozen with ThromboSol and stored so that they may be given back to you if your platelet count drops below a certain level. The frozen platelets can be stored for up to 18 months.

When your platelet count drops below a certain level, you will be scheduled to have a platelet transfusion as part of your standard care.

Before the transfusion you will have blood drawn (around 1-2 teaspoons) to check on the number of platelets in your blood. You will then be randomly assigned (as in the toss of a coin) to either receive the standard platelet transfusion or a ThromboSol-preserved autologous platelet transfusion. After the transfusion, you will have additional blood drawn (around 1-2 teaspoons) to check on the number of platelets in your blood. These procedures will be repeated each time you require a platelet transfusion. However, you will not be randomly assigned again. Each time you receive an additional platelet transfusion, you will be assigned the group different from the one before. The type of transfusions will be alternated. For instance, if you were randomly assigned to receive the frozen platelets for your first transfusion, you will receive the standard transfusion next, then back to the frozen for the third transfusion.

If you develop side effects to the ThromboSol-preserved autologous platelet transfusion or the number of platelets in your blood does not increase after an infusion with the preserved platelets, you will be taken off the study and given a standard platelet transfusion.

This is an investigational study. Up to 54 participants will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1) 1.- Patients in remission with ALL, CLL, AML, CML, MDS will be allowed to participate in this program if their platelet count is >150K, and the hemoglobin level is at least 8.0g/dl. The patient will receive their autologous platelets cryopreserved in ThromboSol or the fresh random platelets (FRP) whenever the need for such transfusions is determined to be clinically indicated by their physician(s).

Exclusion Criteria:

1) Patients with detectable circulating malignant cells or ongoing marrow involvement by the tumor will not be eligible.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Patient Platelet Counts (CCI) Post-transfusion | Baseline and 18-24 hour post-transfusion platelet counts

SECONDARY OUTCOMES:
Patient's Corrected Count Increment (CCI) of autologous transfused platelets stored by cryopreservation with ThromboSol | Platelet counts prior to transfusion and 18-24 hour post-transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lichtiger, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org